CLINICAL TRIAL: NCT00828074
Title: Phase I/II Vinorelbine and Sorafenib as Salvage Therapy in Metastatic Breast Cancer
Brief Title: Sorafenib and Vinorelbine in Treating Women With Stage IV Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08103; P30CA033572 (NIH); CHNMC-08103; BAYER-CHNMC-08103; CDR0000632806 (Registry Identifier: NCI PDQ); NCI-2010-00924 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Sorafenib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (vinorelbine tartrate and sorafenib tosylate) (Experimental): Patients receive sorafenib tosylate PO twice daily on days 1-28 and vinorelbine ditartrate IV on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Drug: vinorelbine ditartrate

INTERVENTIONS:
Drug: sorafenib tosylate — Dose level 1 = 200 mg by mouth two times a day on days 1-28 of a 28 day cycle. Dose level 2 = 200 mg by mouth two times a day on days 1-28 of a 28 day cycle. Dose level 3 = 200 mg by mouth in the am and 400 mg by mouth in the pm on days 1-28 of a 28 day cycle. Dose level 4 = 400 mg by mouth two times a day on days 1-28 of a 28 day cycle.
Drug: vinorelbine ditartrate — Dose level 1 = 20 mg/m2 IV weekly on days 1, 8, and 15 of a 28 day cycle. Dose level 2 = 25 mg/m2 IV weekly on days 1, 8, and 15 of a 28 day cycle. Dose level 3 = 25 mg/m2 IV weekly on days 1, 8, and 15 of a 28 day cycle. Dose level 4 = 25 mg/m2 IV weekly on days 1, 8, and 15 of a 28 day cycle.

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as vinorelbine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sorafenib together with vinorelbine may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of sorafenib when given together with vinorelbine and to see how well they work in treating women with stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety, tolerability, and recommended phase II dose of sorafenib tosylate when administered in combination with vinorelbine ditartrate in women with stage IV adenocarcinoma of the breast. (Phase I)
* To evaluate the 4-month progression-free survival rate in patients treated with this regimen at the maximum tolerated dose. (Phase II)

Secondary

* To determine time to treatment failure in these patients.
* To determine the response rate in these patients.
* To determine the overall survival and progression-free survival of these patients.
* To evaluate the toxicity profile of this regimen.

OUTLINE: This is a phase I, dose-escalation study of sorafenib tosylate followed by a phase II study.

Patients receive oral sorafenib tosylate on days 1-28 and vinorelbine ditartrate IV on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed stage IV adenocarcinoma of the breast; (unless metastatic disease is documented by computed tomography [CT] scan, magnetic resonance imaging [MRI], or bone scan; also, skin disease that has not been biopsied maybe used if in the investigators clinical opinion this represents metastatic disease)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan
* Prior adjuvant therapy, and up to 2 lines of prior chemotherapy (including trastuzumab containing regimens in Her-2 positive patients) for metastatic disease are allowed; prior radiation therapy is allowed, prior hormonal therapy is allowed; the total number of patients enrolled with prior trastuzumab containing regimens will not exceed 10; no more than 50% of enrolled patients will receive the study regimen in a third line setting
* Life expectancy of greater than 6 months
* Performance status: Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2
* Hemoglobin >= 9.0 g/dl
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin =< 1.5 times ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 times the upper limit of normal (ULN) (=< 5 x ULN for patients with liver involvement)
* Creatinine =< 1.5 times ULN
* International normalized ratio (INR) < 1.5 or a prothrombin time (PT)/partial thromboplastin time (PTT) within normal limits; patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate; for patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; women of childbearing potential must have a negative serum pregnancy test performed within 7 days to the start of treatment; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks prior; patients who had bevacizumab within 4 weeks prior to entering the study are allowed
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases are excluded from this clinical trial; patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (> Common Terminology Criteria for Adverse Events [CTCAE] grade 2), symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, cardiac ventricular arrhythmias requiring anti-arrhythmic therapy, or psychiatric illness/social situations that would limit compliance with study requirements
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary hemorrhage/bleeding event >= CTCAE Grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event >= CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug
* Use of St. John's Wort or rifampin (rifampicin)
* Known or suspected allergy to sorafenib or any agent given in the course of this trial
* Pregnant women
* Human immunodeficiency virus (HIV)-positive patients
* Any condition that impairs patient's ability to swallow whole pills
* Any malabsorption problem
* Patients who received prior sunitinib are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thehang H. Luu, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - South Pasadena Cancer Center, Pasadena, California

REFERENCES:
- [Derived] Luu T, Frankel P, Chung C, Chow W, Mortimer J, Hurria A, Somlo G. Phase I/II trial of vinorelbine and sorafenib in metastatic breast cancer. Clin Breast Cancer. 2014 Apr;14(2):94-100. doi: 10.1016/j.clbc.2013.10.013. Epub 2013 Oct 26. PMID 24370210

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I - Vinorelbine at 20mg/m^2; Phase II - Vinorelbine 20mg/m^2: Vinorelbine at 20mg/m^2 weekly intravenous (I.V.) on days 1, 8, 15 and sorafenib 200 mg given orally (p.o.) twice daily for 28 days
- Phase I - Vinorelbine at 25mg/m^2: Vinorelbine at 25mg/m^2 weekly intravenous (I.V.) on days 1, 8, 15 and sorafenib 200 mg given orally (p.o.) twice daily for 28 days
Period: Overall Study
Arm/Group | Phase I - Vinorelbine at 20mg/m^2 | Phase I - Vinorelbine at 25mg/m^2 | Phase II - Vinorelbine 20mg/m^2
Started | 6 | 5 | 35
Completed | 6 | 5 | 35
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1 - Vinorelbine at 20mg/m^2: Vinorelbine at 20mg/m^2 weekly intravenous (I.V.) on days 1, 8, 15 and sorafenib 200 mg given orally (p.o.) twice daily for 28 days
- Dose Level 2 - Vinorelbine at 25mg/m^2: Vinorelbine at 25mg/m^2 weekly intravenous (I.V.) on days 1, 8, 15 and sorafenib 200 mg given orally (p.o.) twice daily for 28 days
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 - Vinorelbine at 20mg/m^2 | Dose Level 2 - Vinorelbine at 25mg/m^2 | Total
Number analyzed (Participants) | 41 | 5 | 46
Age, Continuous [Median (Full Range); unit: years] | 54 [31 to 72] | 59 [46 to 67] | 55 [31 to 72]
Gender [Count of Participants; unit: Participants]
  Female | 41 | 5 | 46
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 5 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Dose Limiting Toxicity in Phase I
Description: Dose Limiting Toxicity (DLT) defined as any treatment-related grade 3 or greater non-hematologic toxicity (excluding alopecia, controllable nausea and vomiting, and serum triglycerides < 1,500 mg/dL which recover within 1 week), grade 4 or greater thrombocytopenia, grade 4 or greater febrile neutropenia requiring hospitalization, or treatment delay of > 2 weeks as a result of unresolved toxicity during the first cycle of therapy.
Time Frame: 4 weeks from start of treatment, up to 2 years
Population: All patients receiving treatment were evaluated for DLT.
Measure: Number; unit: participants with DLTs
Groups:
- Phase I: Dose Level 1 - Vinorelbine at 20mg/m^2: Vinorelbine at 20mg/m^2 weekly intravenous (I.V.) on days 1, 8, 15 and sorafenib 200 mg given orally (p.o.) twice daily for 28 days
- Phase I: Dose Level 2 - Vinorelbine at 25mg/m^2: Vinorelbine at 25mg/m^2 weekly intravenous (I.V.) on days 1, 8, 15 and sorafenib 200 mg given orally (p.o.) twice daily for 28 days
Arm/Group | Phase I: Dose Level 1 - Vinorelbine at 20mg/m^2 | Phase I: Dose Level 2 - Vinorelbine at 25mg/m^2
Number analyzed (Participants) | 6 | 5
participants with DLTs | 0 | 3

2. Primary Outcome: Recommended Phase II Dose
Description: The maximum tolerated dose (MTD) of Vinorelbine is based on toxicities observed during the first cycle and is defined as the highest dose tested in which fewer than 33% of patients experience an attributable DLT to the study drug, when at least 6 patients are treated at that dose and are evaluable for toxicity. Dose escalations proceeded according to a standard 3+3 design.
Time Frame: 4 weeks from start of treatment, up to 2 years
Population: All patients observed for 28 days while receiving a full course of therapy or who experienced a DLT. Patients withdrawing before completion of the first course, for reasons other than DLT, were replaced.
Measure: Number; unit: mg/m^2
Groups:
- Phase I: All patients enrolled on the Phase I (dose-finding) portion of the study.
Arm/Group | Phase I
Number analyzed (Participants) | 11
mg/m^2 | 20

3. Secondary Outcome: Progression-free Survival Rate at 4 Months
Description: Estimated using the product-limit method of Kaplan and Meier.Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 4 months following the last course of treatment
Population: All patients treated at the phase II vinorelbine dose (6 in the phase I portion, 35 in the phase II portion).
Measure: Number; unit: percentage of participants
Groups:
- Dose Level II - Vinorelbine I.V. 20 mg/m^2: Vinorelbine I.V. at 20 mg/m^2 weekly on days 1, 8, 15 and sorafenib at 200 mg given orally twice daily.
Arm/Group | Dose Level II - Vinorelbine I.V. 20 mg/m^2
Number analyzed (Participants) | 41
percentage of participants | 44

4. Secondary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Until disease progression, up to 5 years.
Population: All patients treated at the phase II vinorelbine dose (6 in the phase I portion, 35 in the phase II portion).
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Dose Level II - Vinorelbine 20 mg/m^2: Vinorelbine I.V. at 20 mg/m^2 weekly on days 1, 8, 15 and sorafenib at 200 mg given orally twice daily.
Arm/Group | Dose Level II - Vinorelbine 20 mg/m^2
Number analyzed (Participants) | 41
Months | 4.1 [2.6 to 5.3]

5. Secondary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response Rate defined as percentage of patients achieving a Best Response of either CR or PR.
Time Frame: After 2 cycles of treatment, up to 2 years.
Population: All patients treated at the phase II vinorelbine dose (6 in the phase I portion, 35 in the phase II portion). Patients who complete 2 cycles of treatment or who terminate treatment for reasons of toxicity, or who progress prior to the completion of 2 cycles of therapy on the Phase II portion of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Level II - Vinorelbine 20 mg/m^2
Number analyzed (Participants) | 41
percentage of participants | 10

6. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Until death from any cause, up to 5 years.
Population: All patients treated at the phase II vinorelbine dose (6 in the phase I portion, 35 in the phase II portion).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Level II - Vinorelbine 20 mg/m^2
Number analyzed (Participants) | 41
Months | 15.4 [11.6 to 28.9]

7. Secondary Outcome: Toxicity Profile
Description: Number of Participants with Treatment-Related Grade 3 & 4 Toxicities for Sorafenib and Vinorelbine Combination
Time Frame: 28 days following the last course of treatment
Measure: Number; unit: participants
Groups:
- Phase I & II: Patients receive sorafenib tosylate PO twice daily on days 1-28 and vinorelbine ditartrate IV on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  sorafenib tosylate: Dose level 1 = 200 mg by mouth two times a day on days 1-28 of a 28 day cycle. Dose level 2 = 200 mg by mouth two times a day on days 1-28 of a 28 day cycle.
  vinorelbine ditartrate: Dose level 1 = 20 mg/m2 IV weekly on days 1, 8, and 15 of a 28 day cycle. Dose level 2 = 25 mg/m2 IV weekly on days 1, 8, and 15 of a 28 day cycle.
Arm/Group | Phase I & II
Number analyzed (Participants) | 46
participants
  Anemia | 2
  Leukopenia | 16
  Neutropenia | 16
  Thrombocytopenia | 1
  Alkalosis | 1
  Cellulitis | 1
  Cough | 1
  Diarrhea | 3
  Fatigue | 5
  Genital abscess | 1
  Hand-foot toxicity | 7
  Hiccups | 1
  High glucose level | 1
  Hypertension | 3
  Hypokalemia | 1
  Hyponatremia | 2
  Infection (NOS) | 1
  Low phosphate | 3
  Pulmonary embolus | 1
  Myalgia | 1
  Pain (NOS) | 3
  Phlebitis | 1
  Sensory neuropathy | 1
  Somnolence | 1
  Transaminases/alkaline | 1
  Urinary tract infection | 1

ADVERSE EVENTS:
Time Frame: Adverse Events collected over a period of 22 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Dose Level 1 - Vinorelbine at 20mg/m^2 | Dose Level 2 - Vinorelbine at 25mg/m^2
Serious Adverse Events (participants affected / at risk) | 15/41 | 2/5
Other Adverse Events (participants affected / at risk) | 41/41 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - Vinorelbine at 20mg/m^2 (N=41) | Dose Level 2 - Vinorelbine at 25mg/m^2 (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Coagulopathy (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - Vinorelbine at 20mg/m^2 (N=41) | Dose Level 2 - Vinorelbine at 25mg/m^2 (N=5)
Hemoglobin decreased (Blood and lymphatic system disorders) | 28 (73) | 3 (24)
Lymphatic disorder (Blood and lymphatic system disorders) | 3 (5) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 8 (9) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Endocrine disorder (Endocrine disorders) | 3 (7) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (5) | 1 (2)
Eye disorder (Eye disorders) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 5 (8) | 3 (8)
Watering eyes (Eye disorders) | 2 (5) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 12 (13) | 2 (4)
Constipation (Gastrointestinal disorders) | 15 (22) | 1 (9)
Diarrhea (Gastrointestinal disorders) | 28 (82) | 4 (14)
Dry mouth (Gastrointestinal disorders) | 3 (10) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 6 (8) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 7 (11) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 17 (39) | 3 (6)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (7) | 1 (3)
Nausea (Gastrointestinal disorders) | 21 (42) | 3 (9)
Oral pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 14 (21) | 1 (1)
Chest pain (General disorders) | 3 (4) | 0 (0)
Chills (General disorders) | 6 (9) | 3 (3)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 34 (105) | 4 (18)
Fever (General disorders) | 12 (15) | 1 (1)
General symptom (General disorders) | 3 (4) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 11 (23) | 3 (4)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 2 (4) | 1 (1)
Upper respiratory infection (Infections and infestations) | 5 (8) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 22 (65) | 3 (4)
Alkaline phosphatase increased (Investigations) | 19 (41) | 3 (7)
Aspartate aminotransferase increased (Investigations) | 28 (81) | 5 (17)
Bilirubin increased (Investigations) | 2 (2) | 0 (0)
Coagulopathy (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1) | 1 (3)
Leukocyte count decreased (Investigations) | 35 (100) | 5 (26)
Lymphocyte count decreased (Investigations) | 31 (86) | 2 (13)
Neutrophil count decreased (Investigations) | 30 (83) | 5 (27)
Platelet count decreased (Investigations) | 8 (12) | 0 (0)
Weight loss (Investigations) | 10 (25) | 3 (3)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 18 (44) | 3 (7)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 24 (65) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 13 (27) | 1 (6)
Serum calcium decreased (Metabolism and nutrition disorders) | 13 (22) | 2 (4)
Serum calcium increased (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 6 (9) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 22 (41) | 4 (10)
Serum potassium decreased (Metabolism and nutrition disorders) | 15 (24) | 3 (5)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 20 (38) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (14) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (11) | 5 (11)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 10 (25) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 15 (49) | 3 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (13) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (22) | 2 (4)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 7 (8) | 1 (1)
Headache (Nervous system disorders) | 19 (33) | 2 (3)
Neurological disorder NOS (Nervous system disorders) | 5 (12) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 25 (79) | 1 (3)
Taste alteration (Nervous system disorders) | 10 (28) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 4 (8) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (15) | 0 (0)
Kidney pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (4) | 2 (3)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 5 (7) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (27) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (17) | 0 (0)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 15 (31) | 1 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 6 (17) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 15 (43) | 2 (22)
Dry skin (Skin and subcutaneous tissue disorders) | 13 (36) | 1 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 30 (90) | 4 (33)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (16) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 23 (67) | 1 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 19 (74) | 3 (20)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Sweating (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (3)
Hemorrhage (Vascular disorders) | 3 (8) | 0 (0)
Hot flashes (Vascular disorders) | 7 (17) | 0 (0)
Hypertension (Vascular disorders) | 10 (15) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Vascular disorder (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes